CLINICAL TRIAL: NCT01127672
Title: Platelet Rich Plasma Injection Compared to Corticosteroid Injection for Treatment of Plantar Fasciitis. A Prospective, Randomized Control Trial
Brief Title: Treatment of Plantar Fasciitis With Platelet Rich Plasma
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Principal Investigator, William Bunnell, Medical Doctor, Loma Linda University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 59295
Record Dates: First submitted 2010-05-19; First posted 2010-05-21 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Plantar Fasciitis
Keywords: plantar fasciitis; PRP; platelet rich plasma
MeSH Terms: conditions — Fasciitis, Plantar | interventions — Lidocaine; Adrenal Cortex Hormones

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- control (Active Comparator): corticosteroid injection into the origin of the plantar fascia
  Interventions: Drug: corticosteroid injection
- experimental (Active Comparator): platelet rich plasma injection into the origin of the plantar fascia
  Interventions: Biological: platelet rich plasma

INTERVENTIONS:
Biological: platelet rich plasma — 30 ml of a patient's own blood will be collected via blood draw, maintaining sterile technique. This will then be spun down using a Magellan Autologous Platelet Separator System, yielding platelet rich plasma (PRP).
  Under sterile conditions, patients will receive a 3 cc PRP injection (consisting of their own PRP) with 1 cc of 2% lidocaine into the origin of the plantar fascia, administered by an orthopedic surgeon.
  This will be done using a plantar approach. A peppering technique spreading in clockwise manner will be used to achieve a more expansive zone of delivery, with a maximum of 10 passes through the fascia itself.
  The patient will be monitored for 10 minutes in clinic for adverse reactions.
  Other Names: platelet rich plasma - PRP; xylocaine
  Arms: experimental
Drug: corticosteroid injection — Under sterile conditions, patients will receive a 4 cc injection consisting of 2 cc Celestone Soluspan (6mg/ml) and 2 cc of 1% lidocaine into the origin of the plantar fascia, administered by an orthopedic surgeon.
  This will be done using a plantar approach. A peppering technique spreading in clockwise manner will be used to achieve a more expansive zone of delivery, with a maximum of 10 passes through the fascia itself.
  The patient will be monitored for 10 minutes in clinic for adverse reactions.
  Other Names: betamethasone injectable suspension; xylocaine
  Arms: control

SUMMARY:
The purpose of this investigator-initiated study is to clinically evaluate the efficacy of a new treatment for plantar fasciitis. This treatment consists of a platelet rich plasma injection into the origin of the plantar fascia. It is thought that plasma rich plasma injection will dramatically improve outcomes for patients suffering from plantar fasciitis.

Subjects will be randomized by choosing a slip of paper from an envelope. This process will randomize 25 patients to the experimental group, and 25 patients to the control. The experimental group will undergo a blood draw, allowing for an injection of platelet rich plasma into the origin of the plantar fascia. The control group will undergo a corticosteroid injection into the plantar fascia as the sole treatment. Patients will be followed for three months for pain, and will fill out questionnaires at the initial visit prior to receiving the injection, as well as six and twelve weeks post injection.

These questionnaires will give insight into functionality and pain changes that the plantar fascia is experiencing due to treatment.

Subjects will be outpatients. Subjects may include employees, students, minorities, and elderly, although no subsets of these will be formed.

Subjects will be between 18 and 89 years of age.

In total, subject participation will last approximately 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients presenting with complaints of plantar heel pain, worse with rising in morning and/or after periods of sitting or lying presenting for at least 4 weeks
* Examination reveals maximal tenderness at the attachment of the plantar fascia on the medial tubercle of the calcaneus
* Willingness to participate in an investigational technique
* Willingness to forgo any other concomitant conservative treatment modality; NSAIDS and orthotic devices during the study period

Exclusion Criteria:

* Previous surgery for heel pain
* Nerve related symptoms (radiculopathy, tarsal tunnel syndrome, tarsi sinus syndrome)
* Patient with complex regional pain syndrome
* Achilles tendon pathology
* RA, DM, local or systemic infection, PVD, metabolic disease such as gout, clotting disorder, anticoagulation therapy
* Patients that are pregnant or breastfeeding
* Patients with metastatic cancer
* Dysfunction of the knee, ankle, or foot
* Work related or compensable injury
* Previous treatment: corticosteroid injection in the last 6 months or NSAIDs treatment within the last 7 days

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-05; Primary Completion 2011-05 (Estimated); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Pain and Disability of the Foot and Ankle Through Validated Questionnaires | 15 minutes prior to initial injection of corticosteroid versus platelet rich plasma
  Patients will be asked to fill out 3 questionnaires to provide insight into how their condition is progressing. These questionnaires consist of a visual analog pain score, American Orthopaedic Foot and Ankle Society clinical rating system, and the Foot and Ankle Disability Index. All these questionnaires are externally validated clinical outcome measures that rate foot and ankle pain and dysfunction on various numerical scales. With the exception of the visual analogue scale pain score, there is a direct relationship to the score and positive patient outcome.
Pain and Disability of the Foot and Ankle through Validated Questionnaires | 6 weeks from initial injection of corticosteroid versus platelet rich plasma
  Patients will be asked to fill out 3 questionnaires to provide insight into how their condition is progressing. These questionnaires consist of a visual analog pain score, American Orthopaedic Foot and Ankle Society clinical rating system, and the Foot and Ankle Disability Index. All these questionnaires are externally validated clinical outcome measures that rate foot and ankle pain and dysfunction on various numerical scales. With the exception of the visual analogue scale pain score, there is a direct relationship to the score and positive patient outcome.
Pain and Disability of the Foot and Ankle through Validated Questionnaires | 12 weeks from initial injection of corticosteroid versus platelet rich plasma
  Patients will be asked to fill out 3 questionnaires to provide insight into how their condition is progressing. These questionnaires consist of a visual analog pain score, American Orthopaedic Foot and Ankle Society clinical rating system, and the Foot and Ankle Disability Index. All these questionnaires are externally validated clinical outcome measures that rate foot and ankle pain and dysfunction on various numerical scales. With the exception of the visual analogue scale pain score, there is a direct relationship to the score and positive patient outcome.

CONTACTS AND LOCATIONS:
Overall Officials: William P Bunnell, MD, Principal Investigator — Loma Linda University Department of Orthopaedics
Locations (1):
- Loma Linda University Orthopaedic Center, San Bernadino, California, United States

REFERENCES:
- [Background] League AC. Current concepts review: plantar fasciitis. Foot Ankle Int. 2008 Mar;29(3):358-66. doi: 10.3113/FAI.2008.0358. No abstract available. PMID 18348838
- [Background] Sampson S, Gerhardt M, Mandelbaum B. Platelet rich plasma injection grafts for musculoskeletal injuries: a review. Curr Rev Musculoskelet Med. 2008 Dec;1(3-4):165-74. doi: 10.1007/s12178-008-9032-5. PMID 19468902
- [Background] Lee TG, Ahmad TS. Intralesional autologous blood injection compared to corticosteroid injection for treatment of chronic plantar fasciitis. A prospective, randomized, controlled trial. Foot Ankle Int. 2007 Sep;28(9):984-90. doi: 10.3113/FAI.2007.0984. PMID 17880872
- [Background] Kitaoka HB, Alexander IJ, Adelaar RS, Nunley JA, Myerson MS, Sanders M. Clinical rating systems for the ankle-hindfoot, midfoot, hallux, and lesser toes. Foot Ankle Int. 1994 Jul;15(7):349-53. doi: 10.1177/107110079401500701. PMID 7951968
- [Background] Kon E, Filardo G, Delcogliano M, Presti ML, Russo A, Bondi A, Di Martino A, Cenacchi A, Fornasari PM, Marcacci M. Platelet-rich plasma: new clinical application: a pilot study for treatment of jumper's knee. Injury. 2009 Jun;40(6):598-603. doi: 10.1016/j.injury.2008.11.026. Epub 2009 Apr 19. PMID 19380129
- [Background] Mishra A, Pavelko T. Treatment of chronic elbow tendinosis with buffered platelet-rich plasma. Am J Sports Med. 2006 Nov;34(11):1774-8. doi: 10.1177/0363546506288850. Epub 2006 May 30. PMID 16735582
- [Background] Barrett S, Erredge S. Growth factor for chronic plantar fasciitis. Podiatry Today. 17: 37-42, 2004.